CLINICAL TRIAL: NCT00431067
Title: Phase II Trial of BIBW 2992 in Patients With HER2-positive Metastatic Breast Cancer After Failure of Trastuzumab Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1200.11; 2007-004805-80 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2013-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental): BIBW 2992 (Afatinib) once daily until progression
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992
  Other Names: BIBW 2992 (Afatinib) once daily until progression

SUMMARY:
The primary objective of this trial is to explore the efficacy of BIBW 2992 in HER2 positive metastatic breast cancer patients after failure of trastuzumab containing regimens.

ELIGIBILITY:
Inclusion criteria:

Inclusion Criteria:

1. Male or female patients with confirmed diagnosis of Stage IIIB or IV HER2-positive metastatic breast cancer(HER2 2+ and FISH positive or HER2 3+).
2. Patients must have progressed following receipt of prior standard trastuzumab treatment or standard chemotherapy in conjunction with trastuzumab. Patients with visceral disease or rapid progression should not be included if they have not had previous chemotherapy in addition to trastuzumab. Patients who are intolerant to trastuzumab and who have received adequate chemotherapy and/or hormone therapy are eligible upon progression.
3. Age 18 years or older.
4. Life expectancy of at least four (4) months.
5. Written informed consent that is consistent with ICH-GCP guidelines.
6. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance Score 0, 1 or 2.
7. Patients should not have received treatment with chemotherapy or immune therapy within the last 4 weeks (2 weeks for trastuzumab). Patients should not have received treatment with hormone therapy within the last 2 weeks.
8. Patients must have recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies to CTC less than or equal to Grade 1.
9. Patients must have recovered from previous surgery.
10. Patients must have measurable disease as defined by RECIST criteria.

Exclusion criteria:

Exclusion Criteria:

1. Active infectious disease.
2. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea.
3. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
4. Patients with active/symptomatic brain metastases. Patients with a history of treated brain metastases must have stable or normal MRI scan at screening and be at least three months post-radiation or surgery.
5. Cardiac left ventricular function with resting ejection fraction <50%.
6. Absolute neutrophil count (ANC) less than 1500 cells/mm3.
7. Platelet count less than 100 000 cells/mm3.
8. Bilirubin greater than 1.5 mg/dl (>26 micromol /L, SI unit equivalent).
9. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal.
10. Serum creatinine greater than 1.5 mg/dl (>132 micromol/L, SI unit equivalent).
11. Women and men (and their partners) who are sexually active and unwilling to use a medically acceptable method of contraception.
12. Pregnancy or breast-feeding.
13. Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (including LHRH agonists, or other hormones taken for breast cancer), or participation in another clinical study within the past 4 weeks before start of therapy or concomitantly with this study. Treatment with bisphosphonates is allowed.
14. Prior treatment with an EGFR- or HER2 inhibiting drug (except trastuzumab).
15. Patients unable to comply with the protocol.
16. Active alcohol or drug abuse.
17. Patients with history of other malignancy (except for appropriately treated superficial basal cell skin cancer and surgically cured cervical cancer in situ) unless free of disease for at least 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- United States (6):
  - 1200.11.3 Boehringer Ingelheim Investigational Site, Scottsdale, Arizona
  - 1200.11.7 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 1200.11.4 Boehringer Ingelheim Investigational Site, Santa Monica, California
  - 1200.11.2 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1200.11.1 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.11.5 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
- United Kingdom (6):
  - 1200.11.4401 Boehringer Ingelheim Investigational Site, Bournemouth
  - 1200.11.4402 Boehringer Ingelheim Investigational Site, Crownhill, Plymouth
  - 1200.11.4406 Boehringer Ingelheim Investigational Site, Guildford
  - 1200.11.4405 Boehringer Ingelheim Investigational Site, London
  - 1200.11.4404 Boehringer Ingelheim Investigational Site, Poole
  - 1200.11.4403 Boehringer Ingelheim Investigational Site, Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib 50 mg: Patients received continuous daily dosing with Afatinib 50 mg therapy over 28-day treatment cycles until further disease progression or undue toxicity.
Period: Overall Study
Arm/Group | Afatinib 50 mg
Started | 41 (52 patients screened, 41 treated)
Completed | 0 (On treatment at analysis cut-off date (22-Sep-2009))
Not Completed | 41
Not completed — Other Adverse Event | 9
Not completed — Progressive disease | 30
Not completed — Non-compliance,lost to follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: Objective response (OR) including complete response (CR) and partial response (PR) according to the Response Evaluation Criteria in Solid Tumours (RECIST) criteria .
Time Frame: From first dose of study medication to response measurement, up to 34 month
Population: Treated set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number; unit: Participants
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 41
Participants | 4

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first treatment to the occurrence of tumour progression or death, whichever came first. It was assessed according to RECIST criteria.
Time Frame: From first dose of study medication to the occurrence of progression or death whichever came first, up to 34 month
Population: TS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 41
days | 106 [57 to 117]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first treatment to death or to the last date the patient was known to be alive.
Time Frame: From first dose of study medication to death or to the last date the patient was known to be alive, up to 34 month
Population: TS (14 patients died)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 41
days | 427 [397 to NA] — upper bound can not be calculated due to too few deaths.

4. Secondary Outcome: Time to RECIST Tumour Reponse
Description: The time to OR was the duration from the first treatment to the time when the measurement criteria for CR and/or PR were met according to RECIST criteria.
Time Frame: From first dose of study medication to time when OR measurement was taken.
Population: TS. There were only 4 patients who responded.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 41
days | NA [NA to NA] — Median time of RECIST tumour response was not calculable as there were only 4 patients who responded.

5. Secondary Outcome: Duration of Confirmed OR
Description: Duration of confirmed OR is measured from the time of first OR to the time of progression or death (or date of censoring for progression free survival).
Time Frame: From first OR to time of progression or death
Population: TS - patients with OR only.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Afatinib 50 mg
Number analyzed (Participants) | 4
days | 153.3 (162.2)

ADVERSE EVENTS:
Time Frame: From first dose of study medication to 28 days after study drug discontinuation.
Arm/Group | Afatinib 50 mg
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50 mg (N=41)
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Biliary colic (Hepatobiliary disorders) | 1
Diarrhoea infectious (Infections and infestations) | 1
International normalised ratio decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50 mg (N=41)
Anaemia (Blood and lymphatic system disorders) | 7
Keratoconjunctivitis sicca (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 36
Dry mouth (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Oral pain (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 19
Mucosal inflammation (General disorders) | 5
Pyrexia (General disorders) | 3
Localised infection (Infections and infestations) | 4
Weight decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 27
Skin fissures (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.